CLINICAL TRIAL: NCT02024477
Title: Effect of Saxagliptin (DPP-4 Inhibitor) on Endothelial Progenitor Cells (EPCs) as a Cellular Biomarker for Evaluating Endothelial Dysfunction in Early Type 2 Diabetes Patients
Brief Title: Effect of Saxagliptin on EPCs as a Cellular Biomarker for Evaluating Endothelial Dysfunction in Early T2DM Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Sabyasachi Sen, Associate Professor of Medicine, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV181-305
Record Dates: First submitted 2013-12-13; First posted 2013-12-31 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes
Keywords: endothelial cells; cellular biomarker; endothelial dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo 1 pill daily for 12 weeks
  Interventions: Drug: Placebo
- saxagliptin (Active Comparator): Saxagliptin 5mg once daily for 12 weeks
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — 5 mg tablet once daily for 12 weeks
  Other Names: Onglyza
  Arms: saxagliptin
Drug: Placebo — 1 tablet daily for 12 weeks
  Arms: Placebo

SUMMARY:
Type 2 diabetes is a national epidemic. Diabetes has undesirable effects on blood vessels which may contribute to heart disease. Endothelial Progenitor Cells(EPCs) are found in the blood . Research has shown that improving the survival of these special blood cells may decrease the harmful effects of diabetes on blood vessels and reduce or reverse heart disease. Saxagliptin is an FDA(Food and Drug Administration) approved prescription medicine used along with diet and exercise to lower blood sugar in people with Type 2 diabetes. It is in a class of diabetes medication called DPP-4 inhibitors. DPP-4 inhibitors have been shown to increase EPCs in patients with Type 2 diabetes.

Hypothesis: We believe poor viability and function of EPCs in early diabetes ultimately affects the repair and regeneration of the endothelium and that prompt intervention using saxagliptin with another oral hypoglycemic agent, Metformin, may reduce or reverse cardiovascular risk by improving EPC survival and function above and beyond adequate glucose metabolism control.

DETAILED DESCRIPTION:
Type 2 diabetes is a national epidemic 1,2 with significant macro and microvascular complications. Insulin resistance in prediabetes and early and late diabetes are associated with endothelial dysfunction.

A few studies indicate that EPCs can act as a suitable bio-marker for monitoring cardiovascular morbidity. In this proposal we suggest that EPCs or CD34 positive cells can act as a suitable cellular biomarker for estimating and following endothelial dysfunction in early type 2 diabetes patients.

EPCs have been used as a regenerative tool in ischemic myocardium and diabetic wound healing. Endothelial dysfunction with associated inflammation may be a consequence of excess super-oxide presence in a setting of diabetes which is a pro-oxidative stress condition causing EPC dysfunction and senescence. Therefore monitoring EPC number, function and gene expression may serve as a very useful cellular bio-marker for cardiovascular complications in early type 2 diabetes.

Though lifestyle modification has been proposed as a main stay for prevention and treatment of early type 2 diabetes, several new therapies for diabetes have been developed in recent years. Incretins and incretin mimetics appear to hold promise. Oral DPP-4 inhibitors have been shown to increase EPCs in patients with type 2 diabetes reportedly via SDF-1 alpha up-regulation. Interestingly, up-regulation of SDF-1 alpha and vascular endothelial growth factor (VEGF), both chemotactic factors increase mobilization and recruitment of EPCs in the face of acute ischemic injury for repair and regeneration.

Several studies have shown positive effect of incretins (Glucagon like peptide, GLP-1) and incretin receptor agonists (GLP-1 receptor agonists) on cardiovascular risk factors in type 2 diabetes patients and even in patients with chronic heart failure and left ventricular dysfunction who do not have diabetes.

DPP-4 Inhibitors may have cardio-protective effects of their own, as they increase bio-availability of endogenous GLP-1. They improve blood flow and nitric oxide production in endothelium. These are unique properties not demonstrated by other oral diabetes medications. The mechanism underlying these effects may be mediated by increased nitric oxide bioavailability but is not completely known. It is possible that Saxagliptin, a member of DPP-4 inhibitor group of drugs may be able to improve number and function of CD34+ endothelial progenitor cells by up-regulating chemotactic agent SDF1 alpha (DPP-4 degrades SDF-1) and its receptor CXCR47, 20, 21, 30, 31.

Poor viability and function of EPCs in early diabetes may ultimately affect the repair and regeneration of the endothelium and prompt intervention may reduce or reverse cardiovascular risk by improving EPC survival and function above and beyond adequate glucose metabolism control.

Therefore we would like to explore the effect of saxagliptin in addition to lifestyle intervention, on number and function and gene expression of EPC and impact on endothelial dysfunction in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria

1. Adults aged 40-70 years.
2. Diagnosis of type 2 diabetes within the previous 8 years using criteria of the American Diabetes Association
3. Currently treated with no hypoglycemic agents other than a stable dose (>3 months) of metformin (≥1.0 to ≤2 grams daily).
4. HbA1C between 6 to 9% (both inclusive)
5. BMI 25 to 39.9 kg/m2 (both inclusive)

Exclusion Criteria:

1. Contraindications for moderate exercise
2. Implanted devices (e.g., pacemakers) that may interact with Tanita scale
3. Previous coronary or cerebrovascular event within 6 months of screening or active or clinically significant coronary and/or peripheral vascular disease.
4. Low hematocrit <28 Units
5. Pre-existing liver disease and/or ALT and AST >2.5X's UNL
6. Kidney disease (serum creatinine levels ≥1.5 mg/dL for men, ≥1.4 mg/dL for women,Creatinine Clearance ≤50 mL/min)
7. History of pancreatitis, or cancer (except basal cell carcinoma)
8. Statin use started (or dose change) in the last 3 months.
9. Use of oral or injectable anti-diabetic medication other than Metformin
10. Use of any form of consistent-long term steroid medication (oral, inhaled injected or nasal) within the last 3 months
11. Systolic BP> 140 mmHg and diastolic BP> 90 mmHg
12. Active wounds or recent surgery within 3 months.
13. Inflammatory disease, or current use of anti-inflammatory drugs
14. triglycerides >400 mg/dL
15. untreated hyper/hypothyroidism Additionally, patients who are active smokers, patients who are pregnant, nursing women, and post menopausal women who are on hormone replacement therapy will be excluded.

Patients on low dose oral contraceptives will be allowed to participate as these formulations contain lesser amount of estrogens.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-11; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabyaschi Sen, PhD, MD, Principal Investigator — George Washington University
Locations (1):
- Medical Faculty Associates Inc, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan for sharing IPD with other researchers.

REFERENCES:
- [Derived] Dore FJ, Domingues CC, Ahmadi N, Kundu N, Kropotova Y, Houston S, Rouphael C, Mammadova A, Witkin L, Khiyami A, Amdur RL, Sen S. The synergistic effects of saxagliptin and metformin on CD34+ endothelial progenitor cells in early type 2 diabetes patients: a randomized clinical trial. Cardiovasc Diabetol. 2018 May 3;17(1):65. doi: 10.1186/s12933-018-0709-9. PMID 29724198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from clinic of the Principle Investigator and Sub-Investigators involved in the trial. First patient was recruited on 26 Nov 2013, last patient was recruited on 24 May 2016.
Pre-assignment Details: Screening period lasted 2 weeks. No wash-out or run-in periods were necessary.
Period: Overall Study
Arm/Group | Placebo | Saxagliptin
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Saxagliptin | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (8.5) | 58.3 (5.7) | 57.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 14 | 10 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 13 | 15 | 28
  White | 6 | 5 | 11
  Other | 2 | 1 | 3
Weight [Mean (Standard Deviation); unit: Kg] | 202.3 (38.7) | 202.7 (24.5) | 202.5 (31.6)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.5 (4.8) | 32.3 (4.2) | 31.9 (4.5)
Duration of Diabetes Mellitus II [Mean (Standard Deviation); unit: Years] | 3.5 (1.8) | 3.7 (2.4) | 3.6 (2.1)
HBA1c [Mean (Standard Deviation); unit: mmol/mol] | 6.6 (0.5) | 7.0 (0.8) | 6.8 (0.65)
Fasting Glucose [Mean (Standard Deviation); unit: mg/Dl] | 114.8 (25) | 127.4 (35.9) | 121.1 (30.45)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73] | 93.7 (16.7) | 98.9 (14.5) | 96.3 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: CD34+ Endothelial Progenitor Cells Number
Description: We will use patient's peripheral blood derived CD34+ cells looking at number of CD34+ Endothelial Progenitor Cell as % of the total Mononuclear cell population. Post saxagliptin will be compared to pre saxagliptin measurement
Time Frame: Up to 12 weeks post saxagliptin
Measure: Mean (Standard Deviation); unit: % of Mononuclear Cells
Arm/Group | Placebo | Saxagliptin
Number analyzed (Participants) | 21 | 21
% of Mononuclear Cells | 2.0 (0.3) | 2.8 (0.5)

2. Primary Outcome: CD 34+ Cell Function
Description: function of EPC cell as migration of CD34+ cells in response to SDF-1a ( 100 ng/mL). Results are expressed in fluorescence ratio between cells exposed to the chemotactic factor and cells exposed to chemo attractant-free media ( control) followed by lysis in presence of CyQuant GR dye.
Time Frame: Up to 12 weeks post saxagliptin Up to 12 weeks post saxagliptin: Visit 1 at Baseline, Visit 2 at 6 weeks, and Visit 3 at 12 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | Saxagliptin
Number analyzed (Participants) | 21 | 21
Ratio
  Visit 1 - Week 0 | 1.2 (0.1) | 1.05 (0.06)
  Visit 2 - Week 6 | 1.05 (0.15) | 1.55 (0.2)
  Visit 3 - Week 12 | 1.0 (0.06) | 1.2 (0.05)

3. Secondary Outcome: Serum Endothelial Inflammatory Marker hsCRP
Time Frame: Baseline 6 and 12 weeks post saxagliptin
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Saxagliptin
Number analyzed (Participants) | 21 | 21
mg/L
  Visit 1 - Baseline | 2.4 (0.6) | 2.8 (0.5)
  Visit 2 - Week 6 | 2.9 (0.8) | 2.7 (0.4)
  Visit 3 - Week 12 | 2.9 (0.7) | 2.4 (0.4)

4. Secondary Outcome: Fasting Lipid Profile LDL/HDL
Description: ratio of LDL over HDL
Time Frame: Baseline, 6 and 12 weeks post saxagliptin
Measure: Mean (Standard Deviation); unit: ratio of LDL over HDL
Arm/Group | Placebo | Saxagliptin
Number analyzed (Participants) | 21 | 21
ratio of LDL over HDL
  Visit 1 - Baseline | 2.3 (0.2) | 1.8 (0.1)
  Visit 2 - Week 6 | 2.1 (0.2) | 1.8 (0.1)
  Visit 3 - Week 12 | 2.1 (0.2) | 1.8 (0.2)

5. Secondary Outcome: Glycemic Control
Description: measuring HbA1c levels
Time Frame: Baseline, 6 and 12 weeks post saxagliptin
Measure: Mean (Standard Deviation); unit: % of Glycosylated Hemoglobin
Arm/Group | Placebo | Saxagliptin
Number analyzed (Participants) | 21 | 21
% of Glycosylated Hemoglobin
  Visit 1 - Baseline | 6.6 (0.1) | 7.0 (0.2)
  Visit 2 - Week 6 | 6.6 (0.1) | 6.8 (0.2)
  Visit 3 - Week 12 | 6.5 (0.1) | 6.7 (0.2)

6. Secondary Outcome: Adiposity
Description: measured using a Tanita Body Composition Fat Analyzer scale, measured as percentage body fat
Time Frame: Baseline, 6 and 12 weeks post saxagliptin
Measure: Mean (Standard Deviation); unit: % of Body fat
Arm/Group | Placebo | Saxagliptin
Number analyzed (Participants) | 21 | 21
% of Body fat
  Visit 1 - Baseline | 34 (2) | 37 (2)
  Visit 2 - Week 6 | 34 (2) | 36.5 (2)
  Visit 3 - Week 12 | 35 (2) | 36 (2)

7. Secondary Outcome: Arterial Stiffness
Description: Arterial stiffness assessed using Vascular Flow and wave measurement equipment, SphygmoCor CP system from ATCOR. Reported as Augmentation Index adjusted for a heart rate of 75. Augmentation index (AIx) is a measure of systemic arterial stiffness derived from the ascending aortic pressure waveform. Lower the value, better correlated outcome as positive augmentation represents stiffer artery.
Time Frame: Baseline, 6 and 12 weeks post saxagliptin
Measure: Mean (Standard Deviation); unit: Augmentation Index
Arm/Group | Placebo | Saxagliptin
Number analyzed (Participants) | 21 | 21
Augmentation Index
  Visit 1: Baseline | 18.4 (2.4) | 24.1 (2.1)
  Visit 2: Week 6 | 26 (3.9) | 22.5 (2.0)
  Visit 3: Week 12 | 23.3 (2.3) | 23.1 (2.1)

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: from the day ICF was signed till 1 month after V3.
Arm/Group | Placebo | Saxagliptin
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Saxagliptin (N=21)
Hypertensive Urgency (Cardiac disorders) | 1 | 0
Chest Pain (Cardiac disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Limitations of our study may include the relatively short duration of 12 week Saxagliptin therapy, which may have been inadequate to see significant changes in certain clinical and cellular parameters.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT02024477/Prot_SAP_000.pdf